CLINICAL TRIAL: NCT02615054
Title: Assessment for Long-Term Cardiovascular Impairment Associated With Trastuzumab Cardiotoxicity in HER2-Positive Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-258
Record Dates: First submitted 2015-11-19; First posted 2015-11-25 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Trastuzumab Cardiotoxicity; HER2-Positive Breast Cancer Survivors
Keywords: Cardiovascular Impairment; 15-258
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (3):
- treated with trastuzmab no cardiac effects
  Interventions: Device: 2D Echocardiogram; Device: Cardiopulmonary exercise testing and post-CPET cardiac function
- treated with trastuzmab with cardiac effects
  Interventions: Device: 2D Echocardiogram; Device: Cardiopulmonary exercise testing and post-CPET cardiac function
- healthy volunteers no cancer treatment
  Interventions: Device: 2D Echocardiogram; Device: Cardiopulmonary exercise testing and post-CPET cardiac function

INTERVENTIONS:
Device: 2D Echocardiogram — All patients will undergo a two-dimensional echocardiogram with speckle tracking strain analysis within the MSK echocardiography laboratory.
Device: Cardiopulmonary exercise testing and post-CPET cardiac function — To determine VO2peak, an electronic motorized treadmill test with 12-lead ECG monitoring (Mac ® 5000, GE Healthcare) will be performed by certified exercise physiologists.

SUMMARY:
This is for participants with a history of HER2-positive breast cancer and were treated with chemotherapy that increases the risk of abnormal heart function. Strain (a marker of heart function) is a new method of monitoring heart function in cancer patients and is measured with an ultrasound. Exercise testing is another method that can be used to monitor for abnormal heart function in cancer patients. The purpose of this study is to see if strain and exercise testing can be used to detect for late signs of heart damage from chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Aged ≥ 18 years
* Female
* MSK histologically confirmed primary invasive breast carcinoma
* Pathologically confirmed HER2-positive breast cancer
* Treated with adjuvant trastuzumab (either alone or in combination with other anti-HER2 agents)
* ≥ 2 years since completion of targeted chemotherapy without evidence of disease
* Willing and able to comply with the requirements of the protocol

Patients in the cardiotoxicity (TOX) group must meet the following criteria:

* Development of treatment associated cardiotoxicity during trastuzumab therapy, defined as an absolute decrease from baseline in LVEF by ≥ 10%, to an LVEF of below 55%.
* No clinical signs or symptoms of heart failure (NYHA class III or IV) at the time of cardiotoxicity.

Note: NYHA Class III symptoms include marked limitation of physical activity. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain. NYHA Class IV symptoms include inability to carry on any physical activity without discomfort. Symptoms of heart failure or anginal syndrome may be present at rest, and if any physical activity is undertaken, discomfort is increased.

Patients in the no cardiotoxicity (NO-TOX) group must meet the following criteria:

* Maximum absolute decrease in LVEF ≤ 5% from baseline during trastuzumab therapy.
* Echocardiogram with LVEF assessment performed at baseline (prior to initiation of trastuzumab therapy) and at least two timepoints during trastuzumab therapy.
* LVEF ≥ 55% on each echocardiogram assessment during trastuzumab therapy.
* No clinical signs or symptoms of heart failure (NYHA class III or IV) during trastuzumab treatment.

Note: NYHA Class III symptoms include marked limitation of physical activity. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain. NYHA Class IV symptoms include inability to carry on any physical activity without discomfort. Symptoms of heart failure or anginal syndrome may be present at rest, and if any physical activity is undertaken, discomfort is increased.

Participants in the healthy control group must meet the following criteria:

* Aged ≥ 40 years
* Female
* No history of cancer with the exception of localized basal and/or squamous cell carcinoma of the skin
* No prior history of known cardiac disease (e.g. ischemic heart disease, heart failure, cardiomyopathy, or valvular heart disease [moderate to severe], or significant arrhythmias).
* Willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Inability to provide informed consent
* Presence of metastatic disease
* Treatment with additional cardiotoxic therapy for a secondary malignant neoplasm, or treatment with additional cardiotoxic therapy for breast cancer recurrence since primary breast cancer diagnosis [Note: Patients who are diagnosed with a second primary malignancy are not excluded from participation in the study, unless they meet this exclusion criterion.]
* Subjects must not have any of the following absolute contraindications to cardiopulmonary exercise testing : (a) acute myocardial infarction (within 3-5 days of any planned study procedures), (b) unstable angina, (c) uncontrolled arrhythmias causing symptoms or hemodynamic compromise, (d) symptomatic severe aortic stenosis, (e) recurrent syncope, (f) active endocarditis, (g) acute myocarditis or pericarditis, (h) uncontrolled heart failure, (i) acute pulmonary embolus or pulmonary infarction, (within 3 months of any planned study procedures), (j) thrombosis of lower extremities, (k) suspected dissecting aneurysm, (l) uncontrolled asthma, (m) pulmonary edema (within 3 months of planned study procedures), (n) room air desaturation at rest ≤85%, (o) respiratory failure, (p) acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis), or (q) mental impairment leading to inability to cooperate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potentially eligible subjects who meet the eligibility criteria and who were treated at MSK between 2005 and 2010 will be identified through query of MSK institutional databases. Healthy control subjects will be largely recruited from (though not restricted to) MSK employees.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
cardiac function | 2 years
  Exercise capacity will be assessed by CPET, and echocardiographic images will be obtained immediately after CPET to evaluate contractile reserve.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/